CLINICAL TRIAL: NCT03477162
Title: Metformin Pharmacology in Human Cancers
Brief Title: Metformin Pharmacology in Human Cancers: A Proof of Principle Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment was closed as efforts had become more challenging, and the lab indicated that they were able to obtain their primary objective with the number that had already been enrolled.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Joseph D. Phillips, MD., Staff Physician, Thoracic Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D17188
Record Dates: First submitted 2018-03-14; First posted 2018-03-26 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-11

CONDITIONS: Thoracic Neoplasm
MeSH Terms: conditions — Thoracic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): Patients enrolled will be treated with metformin (administered orally; 750 mg QD for 4 days, then 750 mg BID for 3-6 days; or clinically indicated metformin) for a total of 7-10 days prior to surgery, up until the night before surgery.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be given to patients prior to surgery.

SUMMARY:
This is a presurgical (proof of principle, window of opportunity) study in patients with surgically resectable thoracic tumors to determine steady-state tissue and plasma concentrations of metformin.

DETAILED DESCRIPTION:
To understand the variability in clinical results testing metformin as an anti-cancer agent, it is important to determine the concentrations of metformin that are achievable in tissue. Clinical effects of metformin develop gradually over several days of treatment. Steady-state plasma metformin concentrations are correlated with anti-hyperglycemic response. Thus, achieving steady-state concentrations in this study will allow accurate determination of the most representative concentrations of metformin in normal and cancerous tissues, as well as determine AMP-activated protein kinase (AMPK) signaling differences in these tissues. As tha Primary Objective is to determine the concentration of metformin in tumors, patients will be treated with metformin extended release (ER) (Glucophage® XR), starting at 750 milligrams (mg) oral (PO) once daily (QD) for 4 days, then escalating to 750 mg PO twice daily (BID) for 3-6 days prior to surgery. FDA prescribing information indicates that metformin reaches steady-state plasma concentrations within 24-48 hours after the start of dosing in humans; thus, the 7-to-10-day time frame of this study will allow sufficient time for metformin to reach steady-state plasma concentrations, in addition to time allotted for potential accumulation in tissues. Metformin concentrations will be measured using a validated liquid chromatography-mass spectrometry (LC-MS/MS) assay.

ELIGIBILITY:
Inclusion Criteria:

* Invasive malignant solid tumor of thoracic origin (e.g., lung, esophageal, thymus, mesothelioma, chest wall, mediastinum, trachea, pleura) with the intent to treat or biopsy by surgery as standard of care. Tumor must be ≥2 centimeters (cm).
* Patients with multicentric disease are eligible. Samples from all available tumors are requested for research purposes.
* Patients with Type 2 diabetes mellitus being treated with metformin (any dose) for a clinical indication at the time of study enrollment are eligible, and will continue metformin treatment as clinically indicated during the presurgical study period. Their dose of metformin will NOT be changed.
* Patients not on metformin at the time of study entry must be willing to take metformin extended release (Glucophage® XR, 750 mg QD for 4 days, then 750 mg BID for 3-6 days) for a total of 7-10 days prior to surgery.
* Patients do not require a diagnosis of diabetes to be enrolled in the study.
* All patients must be willing to keep a drug diary indicating the dates and times of metformin administration.

Patients must meet the following clinical laboratory criteria:

* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm3 and platelet count greater than or equal to 75,000/mm3.
* Total bilirubin less than or equal to 1.5x the upper limit of the normal range (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3x ULN.
* Estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73m2 or estimated creatinine clearance (eCrCL) > 60 mL/min
* Ability to give informed consent.
* Patients must be willing to provide 20 milliliters (mL) of blood for research use.
* Patient must be willing to provide consent for use of archived tissue for research.

Exclusion Criteria:

* History of diabetes that is currently being treated without metformin.
* Patients who, at the time of study entry, are not taking metformin for a clinical indication, and who will need a radiographic analysis with an iodinated contrast agent during the metformin study treatment period.
* This criterion does not apply to patients taking clinically indicated metformin at the time of study entry.
* History of liver disease as defined with liver function tests (LFTs) above those in the inclusion
* Known hypersensitivity to metformin.
* History of reactive hypoglycemia.
* Active or history of lactic acidosis, metabolic acidosis, or diabetic ketoacidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Phillips, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Witters LA. The blooming of the French lilac. J Clin Invest. 2001 Oct;108(8):1105-7. doi: 10.1172/JCI14178. No abstract available. PMID 11602616
- [Background] Viollet B, Guigas B, Sanz Garcia N, Leclerc J, Foretz M, Andreelli F. Cellular and molecular mechanisms of metformin: an overview. Clin Sci (Lond). 2012 Mar;122(6):253-70. doi: 10.1042/CS20110386. PMID 22117616
- [Background] Rena G, Pearson ER, Sakamoto K. Molecular mechanism of action of metformin: old or new insights? Diabetologia. 2013 Sep;56(9):1898-906. doi: 10.1007/s00125-013-2991-0. Epub 2013 Jul 9. PMID 23835523
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Background] Gunton JE, Delhanty PJ, Takahashi S, Baxter RC. Metformin rapidly increases insulin receptor activation in human liver and signals preferentially through insulin-receptor substrate-2. J Clin Endocrinol Metab. 2003 Mar;88(3):1323-32. doi: 10.1210/jc.2002-021394. PMID 12629126
- [Background] El-Mir MY, Nogueira V, Fontaine E, Averet N, Rigoulet M, Leverve X. Dimethylbiguanide inhibits cell respiration via an indirect effect targeted on the respiratory chain complex I. J Biol Chem. 2000 Jan 7;275(1):223-8. doi: 10.1074/jbc.275.1.223. PMID 10617608
- [Background] DeFronzo RA, Goodman AM. Efficacy of metformin in patients with non-insulin-dependent diabetes mellitus. The Multicenter Metformin Study Group. N Engl J Med. 1995 Aug 31;333(9):541-9. doi: 10.1056/NEJM199508313330902. PMID 7623902
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Hurst RT, Lee RW. Increased incidence of coronary atherosclerosis in type 2 diabetes mellitus: mechanisms and management. Ann Intern Med. 2003 Nov 18;139(10):824-34. doi: 10.7326/0003-4819-139-10-200311180-00010. PMID 14623620
- [Background] Graham GG, Punt J, Arora M, Day RO, Doogue MP, Duong JK, Furlong TJ, Greenfield JR, Greenup LC, Kirkpatrick CM, Ray JE, Timmins P, Williams KM. Clinical pharmacokinetics of metformin. Clin Pharmacokinet. 2011 Feb;50(2):81-98. doi: 10.2165/11534750-000000000-00000. PMID 21241070
- [Background] Christensen MM, Brasch-Andersen C, Green H, Nielsen F, Damkier P, Beck-Nielsen H, Brosen K. The pharmacogenetics of metformin and its impact on plasma metformin steady-state levels and glycosylated hemoglobin A1c. Pharmacogenet Genomics. 2011 Dec;21(12):837-50. doi: 10.1097/FPC.0b013e32834c0010. PMID 21989078
- [Background] Timmins P, Donahue S, Meeker J, Marathe P. Steady-state pharmacokinetics of a novel extended-release metformin formulation. Clin Pharmacokinet. 2005;44(7):721-9. doi: 10.2165/00003088-200544070-00004. PMID 15966755
- [Background] Shu Y, Sheardown SA, Brown C, Owen RP, Zhang S, Castro RA, Ianculescu AG, Yue L, Lo JC, Burchard EG, Brett CM, Giacomini KM. Effect of genetic variation in the organic cation transporter 1 (OCT1) on metformin action. J Clin Invest. 2007 May;117(5):1422-31. doi: 10.1172/JCI30558. PMID 17476361
- [Background] Tucker GT, Casey C, Phillips PJ, Connor H, Ward JD, Woods HF. Metformin kinetics in healthy subjects and in patients with diabetes mellitus. Br J Clin Pharmacol. 1981 Aug;12(2):235-46. doi: 10.1111/j.1365-2125.1981.tb01206.x. PMID 7306436
- [Background] Giovannucci E, Harlan DM, Archer MC, Bergenstal RM, Gapstur SM, Habel LA, Pollak M, Regensteiner JG, Yee D. Diabetes and cancer: a consensus report. Diabetes Care. 2010 Jul;33(7):1674-85. doi: 10.2337/dc10-0666. PMID 20587728
- [Background] Bodmer M, Meier C, Krahenbuhl S, Jick SS, Meier CR. Long-term metformin use is associated with decreased risk of breast cancer. Diabetes Care. 2010 Jun;33(6):1304-8. doi: 10.2337/dc09-1791. Epub 2010 Mar 18. PMID 20299480
- [Background] Decensi A, Puntoni M, Goodwin P, Cazzaniga M, Gennari A, Bonanni B, Gandini S. Metformin and cancer risk in diabetic patients: a systematic review and meta-analysis. Cancer Prev Res (Phila). 2010 Nov;3(11):1451-61. doi: 10.1158/1940-6207.CAPR-10-0157. Epub 2010 Oct 12. PMID 20947488
- [Background] Evans JM, Donnelly LA, Emslie-Smith AM, Alessi DR, Morris AD. Metformin and reduced risk of cancer in diabetic patients. BMJ. 2005 Jun 4;330(7503):1304-5. doi: 10.1136/bmj.38415.708634.F7. Epub 2005 Apr 22. No abstract available. PMID 15849206
- [Background] Jiralerspong S, Palla SL, Giordano SH, Meric-Bernstam F, Liedtke C, Barnett CM, Hsu L, Hung MC, Hortobagyi GN, Gonzalez-Angulo AM. Metformin and pathologic complete responses to neoadjuvant chemotherapy in diabetic patients with breast cancer. J Clin Oncol. 2009 Jul 10;27(20):3297-302. doi: 10.1200/JCO.2009.19.6410. Epub 2009 Jun 1. PMID 19487376
- [Background] Li D, Yeung SC, Hassan MM, Konopleva M, Abbruzzese JL. Antidiabetic therapies affect risk of pancreatic cancer. Gastroenterology. 2009 Aug;137(2):482-8. doi: 10.1053/j.gastro.2009.04.013. Epub 2009 Apr 16. PMID 19375425
- [Background] Libby G, Donnelly LA, Donnan PT, Alessi DR, Morris AD, Evans JM. New users of metformin are at low risk of incident cancer: a cohort study among people with type 2 diabetes. Diabetes Care. 2009 Sep;32(9):1620-5. doi: 10.2337/dc08-2175. Epub 2009 Jun 29. PMID 19564453
- [Background] Wright JL, Stanford JL. Metformin use and prostate cancer in Caucasian men: results from a population-based case-control study. Cancer Causes Control. 2009 Nov;20(9):1617-22. doi: 10.1007/s10552-009-9407-y. Epub 2009 Aug 4. PMID 19653109
- [Background] Xu H, Aldrich MC, Chen Q, Liu H, Peterson NB, Dai Q, Levy M, Shah A, Han X, Ruan X, Jiang M, Li Y, Julien JS, Warner J, Friedman C, Roden DM, Denny JC. Validating drug repurposing signals using electronic health records: a case study of metformin associated with reduced cancer mortality. J Am Med Inform Assoc. 2015 Jan;22(1):179-91. doi: 10.1136/amiajnl-2014-002649. Epub 2014 Jul 22. PMID 25053577
- [Background] Chae YK, Arya A, Malecek MK, Shin DS, Carneiro B, Chandra S, Kaplan J, Kalyan A, Altman JK, Platanias L, Giles F. Repurposing metformin for cancer treatment: current clinical studies. Oncotarget. 2016 Jun 28;7(26):40767-40780. doi: 10.18632/oncotarget.8194. PMID 27004404
- [Background] Dowling RJ, Zakikhani M, Fantus IG, Pollak M, Sonenberg N. Metformin inhibits mammalian target of rapamycin-dependent translation initiation in breast cancer cells. Cancer Res. 2007 Nov 15;67(22):10804-12. doi: 10.1158/0008-5472.CAN-07-2310. PMID 18006825
- [Background] Mohammed A, Janakiram NB, Brewer M, Ritchie RL, Marya A, Lightfoot S, Steele VE, Rao CV. Antidiabetic Drug Metformin Prevents Progression of Pancreatic Cancer by Targeting in Part Cancer Stem Cells and mTOR Signaling. Transl Oncol. 2013 Dec 1;6(6):649-59. doi: 10.1593/tlo.13556. eCollection 2013 Dec 1. PMID 24466367
- [Background] Zakikhani M, Blouin MJ, Piura E, Pollak MN. Metformin and rapamycin have distinct effects on the AKT pathway and proliferation in breast cancer cells. Breast Cancer Res Treat. 2010 Aug;123(1):271-9. doi: 10.1007/s10549-010-0763-9. Epub 2010 Feb 5. PMID 20135346
- [Background] Jalving M, Gietema JA, Lefrandt JD, de Jong S, Reyners AK, Gans RO, de Vries EG. Metformin: taking away the candy for cancer? Eur J Cancer. 2010 Sep;46(13):2369-80. doi: 10.1016/j.ejca.2010.06.012. Epub 2010 Jul 23. PMID 20656475
- [Background] Poloz Y, Stambolic V. Obesity and cancer, a case for insulin signaling. Cell Death Dis. 2015 Dec 31;6(12):e2037. doi: 10.1038/cddis.2015.381. PMID 26720346
- [Background] Camacho L, Dasgupta A, Jiralerspong S. Metformin in breast cancer - an evolving mystery. Breast Cancer Res. 2015 Jun 26;17(1):88. doi: 10.1186/s13058-015-0598-8. PMID 26111812
- [Background] Dowling RJ, Lam S, Bassi C, Mouaaz S, Aman A, Kiyota T, Al-Awar R, Goodwin PJ, Stambolic V. Metformin Pharmacokinetics in Mouse Tumors: Implications for Human Therapy. Cell Metab. 2016 Apr 12;23(4):567-8. doi: 10.1016/j.cmet.2016.03.006. No abstract available. PMID 27076069
- [Background] Kajbaf F, De Broe ME, Lalau JD. Therapeutic Concentrations of Metformin: A Systematic Review. Clin Pharmacokinet. 2016 Apr;55(4):439-59. doi: 10.1007/s40262-015-0323-x. PMID 26330026
- [Background] Glucophage XR product insert. https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=0ahUKEwjcrMLO8cPXAhWGZiYKHVe1DoMQFggrMAA&url=https%3A%2F%2Fpackageinserts.bms.com%2Fpi%2Fpi_glucophage.pdf&usg=AOvVaw2zAbyMgwlF7wxaXv60vtv3.
- [Background] Lipska KJ, Bailey CJ, Inzucchi SE. Use of metformin in the setting of mild-to-moderate renal insufficiency. Diabetes Care. 2011 Jun;34(6):1431-7. doi: 10.2337/dc10-2361. No abstract available. PMID 21617112
- [Background] Wadamori N, Shinohara R, Ishihara Y. Photoacoustic depth profiling of a skin model for non-invasive glucose measurement. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:5644-7. doi: 10.1109/IEMBS.2008.4650494. PMID 19163997
- [Background] Diabetes Prevention Program Research Group. Long-term safety, tolerability, and weight loss associated with metformin in the Diabetes Prevention Program Outcomes Study. Diabetes Care. 2012 Apr;35(4):731-7. doi: 10.2337/dc11-1299. PMID 22442396
- [Background] Bolen S, Feldman L, Vassy J, Wilson L, Yeh HC, Marinopoulos S, Wiley C, Selvin E, Wilson R, Bass EB, Brancati FL. Systematic review: comparative effectiveness and safety of oral medications for type 2 diabetes mellitus. Ann Intern Med. 2007 Sep 18;147(6):386-99. doi: 10.7326/0003-4819-147-6-200709180-00178. Epub 2007 Jul 16. PMID 17638715

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Patients given Metformin prior to surgery
- Control: Patient not given metformin prior to surgery
Period: Overall Study
Arm/Group | Metformin | Control
Started | 17 | 1
Completed | 14 | 1
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Control | Total
Number analyzed (Participants) | 14 | 1 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (6.0) | 75 | 70.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 1 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 1 | 15
Subject already taking metformin at time of study entry [Count of Participants; unit: Participants] | 13 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Lung Tumor Tissue Concentration of Metformin
Description: To determine the intra-tumor concentrations of metformin, with a standard deviation ≤25% of the mean, in patients with solid tumors of thoracic origin administered metformin extended release.
Time Frame: Within 7 days from surgery
Population: Controls do not receive Metformin and are not included in this analysis.
Measure: Median (Full Range); unit: ng/g
Arm/Group | Metformin
Number analyzed (Participants) | 14
ng/g | 1290 [33 to 4445]

2. Secondary Outcome: Concentration of Metformin in Adipose Tissue
Description: To determine the concentration of metformin in adipose tissue.
Time Frame: Within 7 days from surgery
Measure: Median (Full Range); unit: ng/g
Arm/Group | Metformin
Number analyzed (Participants) | 11
ng/g | 70 [45 to 285]

3. Secondary Outcome: Concentration of Metformin in Tumor-adjacent Normal Tissue
Description: To determine the concentration of metformin in tumor-adjacent normal tissue.
Time Frame: Within 7 days from surgery
Measure: Median (Full Range); unit: ng/g
Arm/Group | Metformin
Number analyzed (Participants) | 12
ng/g | 749 [44 to 3013]

4. Secondary Outcome: Concentration of Metformin in Plasma.
Description: To determine the concentration of metformin in plasma.
Time Frame: Within 7 days from surgery
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Metformin
Number analyzed (Participants) | 12
ng/mL | 450 [18 to 6179]

5. Secondary Outcome: Concentration of Metformin in Whole Blood.
Description: To determine the concentration of metformin in whole blood.
Time Frame: Within 7 days from surgery
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Metformin
Number analyzed (Participants) | 14
ng/mL | 514 [3 to 4238]

6. Other Pre Specified Outcome: AMPK Activity Alterations.
Description: To determine whether metformin alters AMPK activity in tumor cells.
Time Frame: Within 7 days from surgery.
Population: AMPK activities were unable to be evaluated and no data is available.
Arm/Group | Metformin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Events were collected from the time of consent until the day after surgery
Arm/Group | Metformin | Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/1
Other Adverse Events (participants affected / at risk) | 1/14 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=14) | Control (N=1)
diarrhea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT03477162/Prot_SAP_000.pdf